CLINICAL TRIAL: NCT03087487
Title: Real-World Comparative Effectiveness Research and Related Economic Outcomes Among Nonvalvular Atrial Fibrillation Patients Using Oral Anti-coagulants
Brief Title: Clinical and Economic Outcomes of Oral Anticoagulants in Non-valvular Atrial Fibrillation
Acronym: ARISTOPHANES
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-543
Record Dates: First submitted 2017-03-17; First posted 2017-03-22 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Non-Valvular Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- NVAF patients on Warfarin: NVAF patients newly initiated with Warfarin. Non-Interventional.
- NVAF patients on Apixaban: NVAF patients newly initiated on Apixaban. Non-Interventional.
- NVAF patients on Dabigatran: NVAF patients newly initiated with Dabigatran. Non-Interventional.
- NVAF patients on Rivaroxaban: NVAF patients newly initiated with Rivaroxaban. Non-Interventional.

SUMMARY:
The primary objectives of this study are to compare the risk of major bleeding and stroke/systemic embolism (SE) events among oral anticoagulant (OAC)-naïve non-valvular atrial fibrillation (NVAF) patients initiating OAC warfarin or apixaban or dabigatran or rivaroxaban treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Had 1 or more pharmacy claim for apixaban or warfarin or dabigatran or rivaroxaban during the identification period (01-Jan-2013 to 30-Sep-2015). The first OAC pharmacy claim date during the identification period will be designated as the index date
2. Patients 18 years old or older as of the index date
3. At least 1 diagnosis of atrial fibrillation prior to or on index date, identified by any medical claim
4. At least 12 months of baseline period prior to index date with continuous enrollment

Exclusion Criteria:

1. Evidence of valvular heart disease, transient atrial fibrillation, venous thromboembolism during the 12-month baseline period or on the index date
2. Evidence of pregnancy during the study period
3. Had a pharmacy claim for warfarin, apixaban, dabigatran, rivaroxaban, or edoxaban during the 12-month baseline period
4. Had more than 1 oral anticoagulant claim on the index date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NVAF patients who were initiators of warfarin or apixaban or dabigatran or rivaroxaban treatment from 01-Jan-2013 through 30-Sep-2015. All patients who have at least 1 year of baseline data available and no prior OAC use will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 466991 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2023-02-26 (Actual); Study Completion 2023-03-08 (Actual)

PRIMARY OUTCOMES:
Time to first major bleeding event | Up to 33 months
Time to first stroke/systemic embolism (SE) event | Up to 33 months

SECONDARY OUTCOMES:
Major bleeding-related medical costs | Up to 33 months
Stroke/SE-related medical costs | Up to 33 months
All-cause Healthcare costs | Up to 33 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Lip GYH, Keshishian AV, Kang AL, Li X, Dhamane AD, Luo X, Balachander N, Rosenblatt L, Mardekian J, Nadkarni A, Pan X, Di Fusco M, Garcia Reeves AB, Yuce H, Deitelzweig SB. Effectiveness and Safety of Oral Anticoagulants in Patients With Nonvalvular Atrial Fibrillation and Diabetes Mellitus. Mayo Clin Proc. 2020 May;95(5):929-943. doi: 10.1016/j.mayocp.2019.05.032. PMID 32370854
- [Derived] Lip GYH, Keshishian A, Li X, Hamilton M, Masseria C, Gupta K, Luo X, Mardekian J, Friend K, Nadkarni A, Pan X, Baser O, Deitelzweig S. Effectiveness and Safety of Oral Anticoagulants Among Nonvalvular Atrial Fibrillation Patients. Stroke. 2018 Dec;49(12):2933-2944. doi: 10.1161/STROKEAHA.118.020232. PMID 30571400
- [Derived] Li X, Keshishian A, Hamilton M, Horblyuk R, Gupta K, Luo X, Mardekian J, Friend K, Nadkarni A, Pan X, Lip GYH, Deitelzweig S. Apixaban 5 and 2.5 mg twice-daily versus warfarin for stroke prevention in nonvalvular atrial fibrillation patients: Comparative effectiveness and safety evaluated using a propensity-score-matched approach. PLoS One. 2018 Jan 26;13(1):e0191722. doi: 10.1371/journal.pone.0191722. eCollection 2018. PMID 29373602
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm